CLINICAL TRIAL: NCT04753567
Title: nCap Medical Nano-Capacitive Pain Relief Patch vs Placebo, a Prospective Randomized Controlled Trial
Brief Title: nCap Pain Relief Patch vs. Placebo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: nCap Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00127554
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis, Knee
Keywords: pain, arthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Arthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Actual pain patch (Experimental)
  Interventions: Device: nCap pain relief patch
- Sham patch (Placebo Comparator)
  Interventions: Device: Sham Patch

INTERVENTIONS:
Device: nCap pain relief patch — Each participant will be randomly assigned to sham or actual patch. Patches will be worn for 3 weeks. Pain and quality of life will be assessed and compared between groups
  Arms: Actual pain patch
Device: Sham Patch — Sham patch will be worn for 3 weeks exactly like actual pain patch
  Arms: Sham patch

SUMMARY:
The purpose of this study is to determine whether use of the nCap Medical Nano-Capacitive pain relief patch reduces subject pain as measured by subject pain scores, WOMAC scores (pain, stiffness and physical function), global assessment scores, and pain medication change as compared to participants randomly assigned to the sham patch group.

ELIGIBILITY:
Inclusion Criteria:

* Meet Altman's clinical criteria for Knee Osteoarthritis
* Male and Female Adults age 40-79
* VAS pain score of > 4 at the beginning of the study

Exclusion Criteria:

* Subject unable to walk unassisted. Participants must be able to stand/walk for 30 minutes
* Inability to read and understand English. Must be able to complete WOMAC scale and questionnaires
* Severe systemic disease limiting ability to ambulate for 30 minutes
* Use of a TENS unit for one week before study or during study
* History of total knee replacement on the affected knee
* Knee surgery on the affected knee in the last 12 months
* Injection into the knee in the last 6 months
* Knee pain < 411
* Inability to cognitively understand consent form or research study, or inability to give consent
* Diagnosis of fibromyalgia, rheumatoid arthritis, gout, dysplasia, septic arthritis, knee pain from other diseases.
* Malignancy
* Injury to knee within 6 months
* Concomitant use of opioids, NSAIDS or other analgesics for 1 week before trial (or 5 half-lives, whichever is greater)9, or during trial with exception of acetaminophen.
* Pregnant or lactating
* Poor general health (ASA classification of IV+)

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Pain score using VAS scale | After 30 minutes of use
  0-10 pain scale

SECONDARY OUTCOMES:
WOMAC score | 3 weeks
  arthritis assessment score
Sustained pain response | 3 weeks
  0-10 VAS pain score
Global assessment question | 3 weeks
  How the patient feels they are doing
Pain medication monitoring | 3 weeks
  Tylenol use

CONTACTS AND LOCATIONS:
Locations (1):
- Knee Arthritis Clinical Trial Officew, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No